CLINICAL TRIAL: NCT05992259
Title: Auricular Vagus Stimulation and ST-Segment Elevation Myocardial Infarction
Brief Title: Auricular Vagus Stimulation and STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bakulev Scientific Center of Cardiovascular Surgery (Other Government)
Collaborators: State Budget Public Health Institution Scientific Research Institute - Ochapovsky Regional Clinical Hospital (Other Government)
Responsible Party: Principal Investigator, Vladimir A Shvartz, MD, MD, DM, Professor, Bakulev Scientific Center of Cardiovascular Surgery
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #12
Record Dates: First submitted 2023-06-27; First posted 2023-08-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Vagus Nerve Stimulation; Acute Coronary Syndrome; Ischemia Reperfusion Injury
Keywords: auricular stimulation; auricular vagus nerve stimulation; transcutaneous vagus nerve stimulation (TENS); vagus nerve stimulation (VNS); acute coronary syndrome; myocardial ischemia reperfusion injury; ST-segment elevation myocardial infarction; coronary heart disease; acute myocardial infarction; mortality; atrial fibrillation
MeSH Terms: conditions — Acute Coronary Syndrome; Reperfusion Injury; ST Elevation Myocardial Infarction; Coronary Disease; Atrial Fibrillation | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of active stimulation vs. sham stimulation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TENS (Active Comparator): It will be performed attached to the tragus of the left ear.
  Interventions: Device: TENS
- Sham TENS (Sham Comparator): It will be performed attached to the earlobe of the left ear.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — TENS will be performed from the moment of admission to the PCI, during the PCI and for the next 30 minutes after it.

SUMMARY:
At the moment, the invasive strategy for the infarct-associated coronary artery in patients with ST-segment elevation myocardial infarction (STEMI) necessary to save the myocardium and reduce the size of the necrosis zone remains the leading one. However, despite the high efficiency of providing medical care to patients with acute coronary syndrome (ACS), there remains a high mortality and disability of this group of patients. In this regard, the search for new drug and non-drug strategies for the treatment of patients with ACS is actively continuing. Over the past decade, it has been shown that transcutaneous vagus nerve stimulation (TENS) has a cardioprotective effect both in chronic heart failure and in coronary heart disease, improves cardiac function, prevents reperfusion injury, weakens myocardial remodeling, increases the effectiveness of defibrillation and reduces the size of a heart attack. One of the methods of noninvasive stimulation of the afferent fibers of the vagus nerve is percutaneous electrical stimulation of the auricular branch of the vagus nerve. However, further studies are needed to determine whether stimulation of the tragus can improve the long-term clinical outcome in this cohort of patients.

DETAILED DESCRIPTION:
ACS is a combined concept for such life-threatening conditions as acute myocardial infarction (AMI) and unstable angina, which are exacerbations of coronary heart disease. However, despite the high effectiveness of the invasive treatment strategy, there remains a high mortality and disability of this group of patients. One of the reasons for this problem is reperfusion injury of the myocardium during revascularization, since reperfusion itself causes myocardial damage, known as Myocardial Ischemia Reperfusion Injury (MIRI). Every year, new data from experimental studies and small clinical trials appear, confirming the concept that MIRI makes a big contribution to the final size of a heart attack and cardiac myocardial function. Currently, there is no specific treatment aimed at MIRI in patients with STEMI. Thus, new treatment methods are needed that can reduce MIRI in revascularized patients. In the course of small clinical studies, it was shown that against the background of vagus nerve stimulation, a significant decrease in heart rate occurs, inflammatory processes and cellular apoptosis are suppressed, left ventricular remodeling decreases and myocardial contractile function improves. Also, a significant decrease in MIRI is demonstrated with percutaneous stimulation of the vagus nerve in the acute period of myocardial infarction. The data of the first clinical trial with VNS in patients with STEMI were published in 2017 (doi:10.1016/j.jcin.2017.04.036). This experimental study increases the likelihood that this noninvasive therapy can be used to treat patients with STEMI who are undergoing primary percutaneous coronary intervention (PCI). New studies are needed to prove the safety and effectiveness of vagus nerve stimulation in patients with STEMI.

ELIGIBILITY:
Inclusion Criteria:

* patients with STEMI who have signed an informed voluntary consent to participate in the study;
* primary myocardial infarction;
* treatment in the first 12 hours from the onset of pain syndrome;
* primary PCI.

Exclusion Criteria:

* acute heart failure III-IV;
* bradyarrhythmias;
* atrial fibrillation/flutter at the time of switching on;
* Thrombolytic therapy at the prehospital stage;
* a history of myocardial infarction;
* PCI/coronary artery bypass grafting (CABG) in the anamnesis.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality | From date of randomization until the date of death from any cause, assessed up to 14 days.
  The number of patients who died in the hospital.
30-day mortality | From date of randomization until the date of death from any cause, assessed up to 30 days.
  The number of patients who died within 30 days from the development of myocardial infarction.

SECONDARY OUTCOMES:
Number of participants with non-lethal events. | From the date of randomization to the date of any of the listed events, assessed up to 14 days.
  The main hospital non-lethal events (Pulmonary edema, Cardiogenic shock, Cardiac arrhythmias: Atrial fibrillation, Ventricular tachycardia/fibrillation, Accelerated idioventricular rhythm/Atrioventricular block II, III).

OTHER OUTCOMES:
Assessment of the level of myocardial damage. | Diagnosis will be carried out during hospitalization, after 6 hours and on the 4th day of hospitalization.
  Dynamics of Troponin I (hs-cTnI) in blood plasma.
Assessment of the level of inflammation. | Diagnosis will be carried out during hospitalization and after 24 hours.
  Dynamics of high-sensitivity C-reactive protein (hs-CRP) in blood plasma. Dynamics of copeptin (CPP) in blood plasma.
Assessment of the level of heart failure | Diagnosis will be carried out during hospitalization and on the 4th day of hospitalization.
  Dynamics of NT-proBNP in blood plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Shvartz, MD, DM, Principal Investigator — Bakoulev Scientific Center for Cardiovascular Surgery
Locations (1):
- Scientific Research Institute Ochapovsky Regional Clinical Hospital, Krasnodar, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kruchinova S, Gendugova M, Namitokov A, Sokolskaya M, Gilevich I, Tatarintseva Z, Karibova M, Danilov V, Simakin N, Shvartz E, Kosmacheva E, Shvartz V. Low-Frequency Electrical Stimulation of the Auricular Branch of the Vagus Nerve in Patients with ST-Elevation Myocardial Infarction: A Randomized Clinical Trial. J Clin Med. 2025 Mar 10;14(6):1866. doi: 10.3390/jcm14061866. PMID 40142674
- See also: Low-Level Tragus Stimulation for the Treatment of Ischemia and Reperfusion Injury in Patients With ST-Segment Elevation Myocardial Infarction: A Proof-of-Concept Study — https://doi.org/10.1016/j.jcin.2017.04.036
- See also: Vagal Cardioprotection in Reperfused Acute Myocardial Infarction — https://doi.org/10.1016/j.jcin.2017.05.063